CLINICAL TRIAL: NCT02339142
Title: Combined Radiotherapy and Intravenous Steroids for Early Progressive Thyroid Eye Disease
Acronym: CRISEPTED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Peter Dolman, Clinical Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H14-03166
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined radiotherapy and iv corticosteroid (Experimental): Therapy: iv MP 500 mg iv weekly for 6 weeks, then 250 mg iv weekly for 6 weeks
  + External beam radiotherapy: 100 Rads to each orbit x 10 doses
  Interventions: Radiation: External beam radiotherapy; Drug: intravenous corticosteroids (methylprednisolone)
- iv Corticosteroid (Active Comparator): iv MP 500 mg iv weekly for 6 weeks, then 250 mg iv weekly for 6 week No Radiotherapy administered
  Interventions: Drug: intravenous corticosteroids (methylprednisolone)

INTERVENTIONS:
Radiation: External beam radiotherapy — 100 Rads to each lateral orbit x 10 doses
  Arms: Combined radiotherapy and iv corticosteroid
Drug: intravenous corticosteroids (methylprednisolone) — Intravenous methylprednisolone (iv MP) 500 mg weekly x 6 weeks, then iv MP 250 mg x 6 weeks

SUMMARY:
Thyroid eye disease is an autoimmune disorder affecting approximately 50% of individuals with autoimmune thyroid diseases resulting in enlargement of ocular muscles and may lead to congestion of the eyelids and ocular surface, ocular movement restriction and double vision, and optic nerve compression and loss of vision.

First line medical therapy is oral or intravenous corticosteroids (CS), which several studies have shown results in reduction of soft tissue congestion, but some studies suggesting that ocular restriction or visual loss may still occur in spite of CS therapy.i

External beam radiotherapy (XRT) is second line therapy but is controversial, with some studies suggesting benefit in preventing onset of double vision or optic nerve compression while other studies suggest it has no benefit. Most proponents of XRT for TED believe that it is most effective early in the disease evolution. XRT has been shown to be a safe therapy with few side-effects, although retinopathy changes have developed in a small percentage of diabetics and its use is avoided for diabetics.

Combined oral prednisone and XRT has been shown to be more effective in reducing soft tissue inflammation and motility complications than either monotherapy in two different studies.

To date there have been no trials comparing combined XRT and iv CS with iv CS alone for early progressive TED to identify potential benefit in reducing the severity of motility disorders or preventing the onset of dysthyroid optic neuropathy. That is the purpose of this study.

DETAILED DESCRIPTION:
1. Purpose: To demonstrate that combined Radiotherapy (RT) and intravenous corticosteroid (CS) is more effective than iv CS alone in preventing severe motility disruption (including strabismus and primary diplopia) and new-onset dysthyroid optic neuropathy in early progressive thyroid orbitopathy.
2. Hypothesis: Combined RT and iv CS are more effective than iv CS alone in preventing motility problems (reduced field of single binocular vision, reduced ductions, strabismus and worsening diplopia) and in preventing new-onset dysthyroid optic neuropathy in patients with early progressive thyroid orbitopathy.
3. Justification: Standard therapy for progressive TED is iv CS, occasionally supplemented with RT if complications develop in spite of appropriate iv CS therapy. A single retrospective study suggested that early combined treatment may prevent more serious visual complications; this would be the first randomized controlled prospective trial to see if this finding is true.
4. Objectives: Demonstrate a statistically significant reduced rate of new onset optic neuropathy and double vision in patients with progressive TED with combined therapy versus traditional monotherapy.
5. Research Method: Multicentre, institutional based, randomized controlled trial.
6. Statistical Analysis:

Subjects: 100 patients with early progressive TED randomized equally into two groups:

1. Therapy: iv MP 500 mg iv weekly for 6 weeks, then 250 mg iv weekly for 6 weeks

   + XRT 100 Rads to each orbit x 10 doses
2. Control: Same iv MP dose + no XRT

ELIGIBILITY:
Inclusion Criteria:

1. Active TED: Onset less than 6 months AND: Progressive with historic or measured worsening in one or more of VISA parameters in past 2 months: (increasing soft tissue inflammatory changes, development of intermittent or constant diplopia or increased prominence of either eye or lid retraction)
2. Moderately severe TED (all of the following criteria must be met):

V: No optic neuropathy I: Inflammatory score >/= 4/10 S: Intermittent or constant diplopia in any direction except primary gaze AND/OR restriction in ductions to < 30 degrees in any cardinal direction on clinical examination

-

Exclusion Criteria:

1. Age < 35 yrs
2. Diabetes mellitus
3. Previous orbital surgery or radiotherapy for TED
4. Corticosteroid or immunotherapy within previous 2 months for TED
5. Unable or unwilling to provide informed consent-

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
New onset dysthyroid optic neuropathy | 1 year
Progression in ocular motility dysfunction (Improvement or worsening in motility scores and ocular restriction, and need for strabismus surgery) | 1 year
  Improvement or worsening in motility scores and ocular restriction, and need for strabismus surgery at 1 year following initiation of treatment
Participants escaping trial (Number of participants leaving trial because of onset of optic neuropathy or primary strabismus) | 1 year
  Number of participants leaving trial because of onset of optic neuropathy or primary strabismus

SECONDARY OUTCOMES:
VISA inflammatory scores | 6 months and 1 year
  Ocular Inflammatory and congestive scores
Quality of life scores | 6 months and 1 year
  Specific Graves orbitopathy quality of life scoring systems: TED QOL and GO QOL
Proptosis and eyelid retraction changes | 1 year
  Change in proptosis and upper lid retraction
Supplemental iv corticosteroid requirements | 1 year
  Need for additional intravenous corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Dolman, MD, FRCSC, Principal Investigator — University of British Columbia